CLINICAL TRIAL: NCT03515044
Title: A Randomized, Double-Blind, Placebo-Controlled, Dose-Ranging, Multicenter Study to Assess the Efficacy and Safety of Rifaximin Soluble Solid Dispersion (SSD) Tablets Plus Lactulose for the Treatment of Overt Hepatic Encephalopathy (OHE)
Brief Title: Rifaximin Soluble Solid Dispersion (SSD) Tablets Plus Lactulose for the Treatment of Overt Hepatic Encephalopathy (OHE)
Acronym: OHE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bausch Health Americas, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RNHE2041
Record Dates: First submitted 2018-04-12; First posted 2018-05-03 (Actual); Results first posted 2023-04-13 (Actual); Last update posted 2023-04-13 (Actual); Status verified 2023-03

CONDITIONS: Overt Hepatic Encephalopathy

STUDY DESIGN:
Intervention Model Description: Randomized, Double-Blind, Placebo-Controlled, Dose-Ranging, Multicenter Study
Who Masked: Participant, Care Provider, Investigator
Masking Description: Blinding will be maintained in the QD SSD cohorts by administering placebo as the second daily dose.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Cohort 1 40 mg Rifaximin SSD once daily (Experimental): 40 mg Rifaximin immediate release (IR) rifaximin SSD once daily (QD) and lactulose
  Interventions: Drug: 40 mg Rifaximin SSD once daily
- Cohort 2 40 mg Rifaximin SSD twice daily (Experimental): 40 mg Rifaximin immediate release (IR) rifaximin SSD twice daily (BID) and lactulose
  Interventions: Drug: 40 mg Rifaximin SSD twice daily
- Cohort 3 80 mg Rifaximin SSD once daily (Experimental): 80 mg Rifaximin sustained extended release (SER) rifaximin SSD once daily (QD) and lactulose
  Interventions: Drug: 80 mg Rifaximin SSD once daily
- Cohort 4 80 mg Rifaximin SSD twice daiy (Experimental): 80 mg Rifaximin sustained extended release (SER) rifaximin SSD twice daily (BID) and lactulose
  Interventions: Drug: 80 mg Rifaximin SSD twice daily
- Cohort 5 Placebo twice daily (Experimental): SSD placebo twice daily (BID) and lactulose
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: 40 mg Rifaximin SSD once daily — SSD once daily (QD)
  Arms: Cohort 1 40 mg Rifaximin SSD once daily
Drug: 40 mg Rifaximin SSD twice daily — SSD twice daily (BID)
  Arms: Cohort 2 40 mg Rifaximin SSD twice daily
Drug: 80 mg Rifaximin SSD once daily — SSD once daily (QD)
  Arms: Cohort 3 80 mg Rifaximin SSD once daily
Drug: 80 mg Rifaximin SSD twice daily — SSD twice daily (BID)
  Arms: Cohort 4 80 mg Rifaximin SSD twice daiy
Drug: Placebo — Administered twice daily (BID)
  Arms: Cohort 5 Placebo twice daily

SUMMARY:
Study to Assess the Efficacy and Safety of Rifaximin Soluble Solid Dispersion (SSD) Tablets Plus Lactulose for the Treatment of Overt Hepatic Encephalopathy (OHE).

DETAILED DESCRIPTION:
The primary objective of this study is to assess the efficacy of rifaximin SSD plus lactulose versus placebo plus lactulose for the treatment of overt hepatic encephalopathy (OHE). The secondary objectives of this study are to assess the safety of rifaximin SSD in subjects with OHE and to assess the effects of treatment with rifaximin SSD on key secondary endpoints.

ELIGIBILITY:
Inclusion Criteria:

* Male or female age 18 to 75 years of age (inclusive) at the time of screening.
* Females of childbearing potential, defined as a female who is fertile following menarche, must have a negative serum pregnancy test at screening and agree to use an acceptable method of contraception throughout their participation in the study.

Note: Female subjects who have been surgically sterilized (e.g., hysterectomy or bilateral tubal ligation) or who are postmenopausal (defined as total cessation of menses for > 1 year) will not be considered "female subjects of childbearing potential".

* Subject is hospitalized with liver cirrhosis and/or OHE and has a confirmed diagnosis of OHE at Baseline.
* Subject has a Grade 2 or Grade 3 HE episode according to the HE Grading Instrument (HEGI) following 8 to 12 hours of intravenous (IV) hydration and lactulose treatment.

Exclusion Criteria:

* Subject has an uncontrolled major psychiatric disorder including major depression or psychoses as determined by the investigator.
* Subject has been diagnosed with an infection for which they are currently taking oral or parenteral antibiotics, which cannot be discontinued at time of enrollment. Note: Subjects currently taking Rifaximin are not excluded
* Subject shows presence of intestinal obstruction or has inflammatory bowel disease.
* Subject has uncontrolled Type 1 or Type 2 diabetes. Note: Subjects with controlled diabetes may be enrolled if they are on stable doses of oral hypoglycemic drugs for at least 3 months prior to screening, and demonstrate clinically acceptable blood glucose control at Baseline, as determined by the investigator.
* Subject has an active malignancy (exceptions: non-melanoma skin cancers).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2018-09-13 (Actual); Primary Completion 2020-03-12 (Actual); Study Completion 2020-03-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Angela Bulawski, Study Director — Bausch Health
Locations (34):
- United States (34):
  - Bausch Health Site 18, Corona del Mar, California
  - Bausch Health Site 15, Los Angeles, California
  - Bausch Health Site 19, Los Angeles, California
  - Bausch Health Site 04, San Francisco, California
  - Bausch Health Site 13, Bristol, Connecticut
  - Bausch Health Site 08, Miami, Florida
  - Bausch Health Site 05, Chicago, Illinois
  - Bausch Health Site 33, Iowa City, Iowa
  - Bausch Health Site 03, Boston, Massachusetts
  - Bausch Health Site 07, Detroit, Michigan
  - Bausch Health 01, Detroit, Michigan
  - Bausch Health Site 25, Tupelo, Mississippi
  - Bausch Health Site 24, St Louis, Missouri
  - Bausch Health Site 27, Newark, New Jersey
  - Bausch Health Site 36, Brooklyn, New York
  - Bausch Health Site 09, New York, New York
  - Bausch Health Site 28, New York, New York
  - Bausch Health Site 17, Cincinnati, Ohio
  - Bausch Health Site 23, Columbus, Ohio
  - Bausch Health Site 11, Philadelphia, Pennsylvania
  - Bausch Health Site 26, Philadelphia, Pennsylvania
  - Bausch Health Site 10, Philadelphia, Pennsylvania
  - Bausch Health Site 12, Pittsburgh, Pennsylvania
  - Bausch Health Site 16, Charleston, South Carolina
  - Bausch Health Site 22, Dallas, Texas
  - Bausch Health Site 35, Dallas, Texas
  - Bausch Health Site 31, Dallas, Texas
  - Bausch Health Site 02, Houston, Texas
  - Bausch Health Site 37, Houston, Texas
  - Bausch Health Site 30, Richmond, Virginia
  - Bausch Health Site 06, Richmond, Virginia
  - Bausch Health Site 21, Seattle, Washington
  - Bausch Health Site 14, Seattle, Washington
  - Bausch Health Site 20, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Bajaj JS, Hassanein TI, Pyrsopoulos NT, Sanyal AJ, Rahimi RS, Heimanson Z, Israel RJ, Rockey DC. Dosing of Rifaximin Soluble Solid Dispersion Tablets in Adults With Cirrhosis: 2 Randomized, Placebo-controlled Trials. Clin Gastroenterol Hepatol. 2023 Mar;21(3):723-731.e9. doi: 10.1016/j.cgh.2022.05.042. Epub 2022 Jun 22. PMID 35750249

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were randomized into 5 possible double-blind treatment arms during the Double-Blind Period. Upon completion of the Double-Blind Period, participants could continue in the 30 day Open-Label Extension Period in which all participants received rifaximin 550 mg.
Groups:
- Cohort 1 40 mg Rifaximin SSD Once Daily: 40 mg Rifaximin immediate release (IR) rifaximin SSD once daily (QD) and lactulose
  40 mg Rifaximin SSD once daily: SSD once daily (QD) and lactulose
  lactulose: to be taken in the recommended adult size dosage.
- Cohort 2 40 mg Rifaximin SSD Twice Daily: 40 mg Rifaximin immediate release (IR) rifaximin SSD twice daily (BID) and lactulose
  40 mg Rifaximin SSD twice daily: SSD twice daily (BID) and lactulose
  lactulose: to be taken in the recommended adult size dosage.
- Cohort 3 80 mg Rifaximin SSD Once Daily: 80 mg Rifaximin sustained extended release (SER) rifaximin SSD once daily (QD) and lactulose
  80 mg Rifaximin SSD once daily: SSD once daily (QD) and lactulose
  lactulose: to be taken in the recommended adult size dosage.
- Cohort 4 80 mg Rifaximin SSD Twice Daiy: Cohort 4 80 mg Rifaximin SSD twice daily (BID) and lactulose
  80 mg Rifaximin SSD twice daily: SSD twice daily (BID) and lactulose
  lactulose: to be taken in the recommended adult size dosage.
- Cohort 5 Placebo Twice Daily: SSD placebo twice daily (BID) and lactulose
  Placebo: Administered twice daily (BID) and lactulose
  lactulose: to be taken in the recommended adult size dosage.
- Open-Label Rifaximin 550 mg: After completion of the Double-Blind Period, participants could continue in the 30 day Open-Label Extension Period
Period: Double-Blind Period
Arm/Group | Cohort 1 40 mg Rifaximin SSD Once Daily | Cohort 2 40 mg Rifaximin SSD Twice Daily | Cohort 3 80 mg Rifaximin SSD Once Daily | Cohort 4 80 mg Rifaximin SSD Twice Daiy | Cohort 5 Placebo Twice Daily | Open-Label Rifaximin 550 mg
Started | 15 | 15 | 14 | 13 | 14 | 0
Completed | 13 | 13 | 8 | 11 | 8 | 0
Not Completed | 2 | 2 | 6 | 2 | 6 | 0
Period: Open-label Extension Period
Arm/Group | Cohort 1 40 mg Rifaximin SSD Once Daily | Cohort 2 40 mg Rifaximin SSD Twice Daily | Cohort 3 80 mg Rifaximin SSD Once Daily | Cohort 4 80 mg Rifaximin SSD Twice Daiy | Cohort 5 Placebo Twice Daily | Open-Label Rifaximin 550 mg
Started | 0 | 0 | 0 | 0 | 0 | 53
Completed | 0 | 0 | 0 | 0 | 0 | 31
Not Completed | 0 | 0 | 0 | 0 | 0 | 22

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 40 mg Rifaximin SSD Once Daily | Cohort 2 40 mg Rifaximin SSD Twice Daily | Cohort 3 80 mg Rifaximin SSD Once Daily | Cohort 4 80 mg Rifaximin SSD Twice Daiy | Cohort 5 Placebo Twice Daily | Total
Number analyzed (Participants) | 15 | 15 | 14 | 13 | 14 | 71
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.3 (14.88) | 61.1 (8.02) | 63.0 (7.94) | 61.8 (8.07) | 60.0 (9.25) | 61.4 (9.84)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 7 | 9 | 8 | 2 | 33
  Male | 8 | 8 | 5 | 5 | 12 | 38
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 3 | 0 | 2 | 3 | 2 | 10
  White | 12 | 13 | 12 | 10 | 9 | 56
  More than one race | 0 | 1 | 0 | 0 | 2 | 3
  Unknown or Not Reported | 0 | 1 | 0 | 0 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Time to Overt Hepatic Encephalopathy (OHE) Resolution Determined Using the Hepatic Encephalopathy Grading Instrument (HEGI), Defined as HEGI Score < 2
Description: A participant was considered to have an overt HE episode if at least one of the following applied: (1) Disorientated to time or place or person, (2) Lethargic and has asterixis, (3) Inability to assess the patient due to disorientation to time and place and person; and/or somnolence, and/or coma. Severity of OHE episodes was graded using the HEGI scale, where Grade 1 is no clinical findings of OHE, and Grade 4 is comatose. Higher scores on the scale have higher severity (worse outcome).
Time Frame: 14 days
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | Cohort 1 40 mg Rifaximin SSD Once Daily | Cohort 2 40 mg Rifaximin SSD Twice Daily | Cohort 3 80 mg Rifaximin SSD Once Daily | Cohort 4 80 mg Rifaximin SSD Twice Daiy | Cohort 5 Placebo Twice Daily
Number analyzed (Participants) | 15 | 15 | 14 | 13 | 14
hours | 36.1 [12.07 to 63.50] | 21.1 [13.05 to 47.68] | 45.9 [22.75 to 80.37] | 17.9 [11.68 to 58.75] | 62.7 [20.00 to 168.88]

2. Secondary Outcome: Time to Improvement in Hepatic Encephalopathy Grading Instrument (HEGI) Score, Defined as at Least One Grade Decrease (Improvement)
Description: as for outcome 1
Time Frame: 14 days
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Cohort 1 40 mg Rifaximin SSD Once Daily | Cohort 2 40 mg Rifaximin SSD Twice Daily | Cohort 3 80 mg Rifaximin SSD Once Daily | Cohort 4 80 mg Rifaximin SSD Twice Daiy | Cohort 5 Placebo Twice Daily
Number analyzed (Participants) | 15 | 15 | 14 | 13 | 14
days | 2.5 [2.00 to 4.00] | 2.0 [NA to NA] — Confidence intervals could not be calculated for Cohort 2, due to lack of variation in the time to event. | 2.0 [2.00 to 4.00] | 2.0 [2.00 to 4.00] | 3.0 [2.00 to 8.00]

3. Secondary Outcome: Time to Hospital Discharge
Description: Time in days until discharge from the hospital
Time Frame: 14 days
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Cohort 1 40 mg Rifaximin SSD Once Daily | Cohort 2 40 mg Rifaximin SSD Twice Daily | Cohort 3 80 mg Rifaximin SSD Once Daily | Cohort 4 80 mg Rifaximin SSD Twice Daiy | Cohort 5 Placebo Twice Daily
Number analyzed (Participants) | 15 | 15 | 14 | 13 | 14
days | 3.0 [2.00 to 4.00] | 3.0 [2.00 to 4.00] | 3.0 [2.00 to 4.00] | 4.0 [3.00 to 4.00] | 4.5 [2.00 to 6.00]

ADVERSE EVENTS:
Time Frame: Participants were randomized into 5 possible double-blind treatment arms (Cohorts 1 to 5) during the Double-Blind Period, in which adverse events were assessed up to 14 days. Upon completion of the Double-Blind Period, participants could continue in the 30 day Open-Label Extension Period in which all participants received rifaximin 550 mg. Adverse events were monitored/assessed up to a total of 44 days.
Arm/Group | Cohort 1 40 mg Rifaximin SSD Once Daily | Cohort 2 40 mg Rifaximin SSD Twice Daily | Cohort 3 80 mg Rifaximin SSD Once Daily | Cohort 4 80 mg Rifaximin SSD Twice Daiy | Cohort 5 Placebo Twice Daily | Open-label Rifaximin 550 mg
All-Cause Mortality (participants affected / at risk) | 2/15 | 0/15 | 2/14 | 1/13 | 1/14 | 13/53
Serious Adverse Events (participants affected / at risk) | 3/15 | 1/15 | 3/14 | 1/13 | 2/14 | 33/53
Other Adverse Events (participants affected / at risk) | 2/15 | 3/15 | 4/14 | 5/13 | 3/14 | 5/53
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 40 mg Rifaximin SSD Once Daily (N=15) | Cohort 2 40 mg Rifaximin SSD Twice Daily (N=15) | Cohort 3 80 mg Rifaximin SSD Once Daily (N=14) | Cohort 4 80 mg Rifaximin SSD Twice Daiy (N=13) | Cohort 5 Placebo Twice Daily (N=14) | Open-label Rifaximin 550 mg (N=53)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Angina pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac distress (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal Pain Upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abominal Pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 2 (2)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Multiple organ dysfunction syndrome (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chronic hepatic failure (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cirrhosis alcoholic (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hepatic cirrhosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hepatorenal syndrome (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Bacteremia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Kidney infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Peritonitis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Septic shock (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Staphylococcal bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Accidental overdose (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyochloraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cerebral artery embolism (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hepatic encephalopathy (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 13 (13)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (5)
Mental status changes (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 40 mg Rifaximin SSD Once Daily (N=15) | Cohort 2 40 mg Rifaximin SSD Twice Daily (N=15) | Cohort 3 80 mg Rifaximin SSD Once Daily (N=14) | Cohort 4 80 mg Rifaximin SSD Twice Daiy (N=13) | Cohort 5 Placebo Twice Daily (N=14) | Open-label Rifaximin 550 mg (N=53)
Arrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Eye disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Umbilical hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hepatorenal syndrome (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Clostridium difficile (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinusitis fungal (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypernatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dementia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatic encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Contact sponsor for details.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-01-08): https://cdn.clinicaltrials.gov/large-docs/44/NCT03515044/Prot_SAP_000.pdf